CLINICAL TRIAL: NCT01802580
Title: Using an Internet Study to Improve Adherence for Psoriasis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00021783
Record Dates: First submitted 2013-02-20; First posted 2013-03-01 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Fluocinonide; Ointments

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention - internet reminder survey (Experimental): Treatment phase is 12 months. During the intervention, each subject will receive fluocinonide 0.05% ointment, a standard treatment for psoriasis. If their psoriasis could be suitably treated with fluocinonide, then they will be asked to participate in the study. At the initial study visit, fluocinonide will be dispensed in a small jar with a MEMS® electronic monitoring cap attached. Subjects will be asked to apply the medication twice daily. They will be asked to the entire affected area, excluding face and genitals. Subjects will be instructed to apply the smallest amount of study medication sufficient to cover the affected areas. At the end of the treatment phase, subjects will have a feedback session with specific results of adherence behavior revealed. They will receive weekly surveys via internet to complete.
  Interventions: Behavioral: Internet Survey; Drug: fluocinonide 0.05% ointment
- Standard of care, no internet survey (Experimental): Standard treatment for psoriasis. If it is felt that their psoriasis could be suitably treated with fluocinonide, then they will be asked to participate in the study. At the initial study visit, fluocinonide will be dispensed to the subjects in a small jar with a MEMS® electronic monitoring cap attached. Subjects will be asked to apply the medication twice daily. All subjects will be assigned to treatment with topical fluocinonide to the entire affected area, excluding face and genitals. Subjects will be instructed to apply the smallest amount of study medication sufficient to cover the affected areas. At the end of the treatment phase, subjects will have a feedback session with specific results of adherence behavior revealed.
  Interventions: Drug: fluocinonide 0.05% ointment

INTERVENTIONS:
Behavioral: Internet Survey
  Arms: Intervention - internet reminder survey
Drug: fluocinonide 0.05% ointment
  Other Names: Fluonex; Lonide; Lyderm; Fluocinonide-E; Lidex; Lidex-E; Vanos; Licon; Dermacin; Fluex

SUMMARY:
To evaluate whether participation in an Internet-based intervention helps improve short-term and long-term psoriasis treatment outcomes, in particular, adherence.

DETAILED DESCRIPTION:
An investigator-blinded, prospective study of subjects with mild to moderate psoriasis will be conducted. Forty subjects ages 18 years and older will be enrolled.The Internet-based survey will be piloted to evaluate its effect on adherence to topical psoriasis medication. Subjects randomized in a 1:1 ratio to the Internet-survey group will log their impression of the state of their psoriasis on a weekly basis. Subjects in both the intervention and control groups will receive standard-of-care topical fluocinonide 0.05% ointment to be applied to affected areas on the skin twice daily. Adherence to fluocinonide will be assessed using Medication Event Monitoring System (MEMS®) caps, electronic monitors affixed to the medication containers. Investigators and subjects will be blinded to the adherence data until the final (Month 12) treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 18 years or older of age with a diagnosis of mild to moderate psoriasis by a dermatologist will be eligible for participation.
* Less than 20% of body surface involvement for psoriasis.
* Subject is capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* The subject is able to complete the study and comply with study instructions, including attending all study visits.
* In general good health with no other skin disease, disease state or physical condition which would impair evaluation of psoriasis or which would increase health risk by study participation

Exclusion Criteria:

* Individuals younger than 18 years of age.
* Known allergy or sensitivity to topical fluocinonide.
* Inability to complete all study-related visits, or inability to complete the Internet survey due to inadequate Internet access.
* Introduction of any other prescription medication, topical or systemic, for psoriasis while participating in the study. Subjects who are on systemic anti-inflammatory treatments for psoriasis must be on a stable dose for at least 3 months prior to enrollment.
* Any skin condition or disease that may require concurrent therapy or may confound evaluations
* Current enrollment in any research study involving an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Camisa C. Psoriasis. Oxford: Blackwell Scientiﬁc Publications, 1994
- [Background] Piacquadio D, Kligman A. The critical role of the vehicle to therapeutic efficacy and patient compliance. J Am Acad Dermatol. 1998 Aug;39(2 Pt 3):S67-73. doi: 10.1016/s0190-9622(98)70448-7. No abstract available. PMID 9703127
- [Background] Witkowski JA. Compliance: the dermatologic patient. Int J Dermatol. 1988 Nov;27(9):608-11. doi: 10.1111/j.1365-4362.1988.tb02416.x. No abstract available. PMID 3068168
- [Background] Richards HL, Fortune DG, O'Sullivan TM, Main CJ, Griffiths CE. Patients with psoriasis and their compliance with medication. J Am Acad Dermatol. 1999 Oct;41(4):581-3. PMID 10495380
- [Background] Fouere S, Adjadj L, Pawin H. How patients experience psoriasis: results from a European survey. J Eur Acad Dermatol Venereol. 2005 Nov;19 Suppl 3:2-6. doi: 10.1111/j.1468-3083.2005.01329.x. PMID 16274404
- [Background] van de Kerkhof PC, de Hoop D, de Korte J, Cobelens SA, Kuipers MV. Patient compliance and disease management in the treatment of psoriasis in the Netherlands. Dermatology. 2000;200(4):292-8. doi: 10.1159/000018390. PMID 10894958
- [Background] Carroll CL, Feldman SR, Camacho FT, Manuel JC, Balkrishnan R. Adherence to topical therapy decreases during the course of an 8-week psoriasis clinical trial: commonly used methods of measuring adherence to topical therapy overestimate actual use. J Am Acad Dermatol. 2004 Aug;51(2):212-6. doi: 10.1016/j.jaad.2004.01.052. PMID 15280839
- [Background] Yentzer BA, Wood AA, Sagransky MJ, O'Neill JL, Clark AR, Williams LL, Feldman SR. An Internet-based survey and improvement of acne treatment outcomes. Arch Dermatol. 2011 Oct;147(10):1223-4. doi: 10.1001/archdermatol.2011.277. No abstract available. PMID 22006146
- [Background] Zaghloul SS, Goodfield MJ. Objective assessment of compliance with psoriasis treatment. Arch Dermatol. 2004 Apr;140(4):408-14. doi: 10.1001/archderm.140.4.408. PMID 15096368
- [Background] Zschocke I, Mrowietz U, Karakasili E, Reich K. Non-adherence and measures to improve adherence in the topical treatment of psoriasis. J Eur Acad Dermatol Venereol. 2014 May;28 Suppl 2:4-9. doi: 10.1111/jdv.12445. PMID 24684738
- [Background] Laufs U, Bohm M, Kroemer HK, Schussel K, Griese N, Schulz M. [Strategies to improve medication adherence]. Dtsch Med Wochenschr. 2011 Aug;136(31-32):1616-21. doi: 10.1055/s-0031-1281566. Epub 2011 Aug 1. German. PMID 21809255
- [Background] McGrady ME, Hommel KA. Medication adherence and health care utilization in pediatric chronic illness: a systematic review. Pediatrics. 2013 Oct;132(4):730-40. doi: 10.1542/peds.2013-1451. Epub 2013 Sep 2. PMID 23999953
- [Background] Storm A, Andersen SE, Benfeldt E, Serup J. One in 3 prescriptions are never redeemed: primary nonadherence in an outpatient clinic. J Am Acad Dermatol. 2008 Jul;59(1):27-33. doi: 10.1016/j.jaad.2008.03.045. Epub 2008 May 7. PMID 18467003
- [Background] Aslam I, Feldman SR. Practical Strategies to Improve Patient Adherence to Treatment Regimens. South Med J. 2015 Jun;108(6):325-31. doi: 10.14423/SMJ.0000000000000294. No abstract available. PMID 26079456
- [Background] Feldman SR. Practical Ways to Improve Patients' Treatment Outcomes. Winston-Salem, NC:Medical Quality Enhancement Corporation, 2008.
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Helping People Change, 3rd edn. New York: Guilford Press, 2013.
- [Background] van der Meer V, van den Hout WB, Bakker MJ, Rabe KF, Sterk PJ, Assendelft WJ, Kievit J, Sont JK; SMASHING (Self-Management in Asthma Supported by Hospitals, ICT, Nurses and General Practitioners) Study Group. Cost-effectiveness of Internet-based self-management compared with usual care in asthma. PLoS One. 2011;6(11):e27108. doi: 10.1371/journal.pone.0027108. Epub 2011 Nov 11. PMID 22096523
- [Background] Feinstein AR. On white-coat effects and the electronic monitoring of compliance. Arch Intern Med. 1990 Jul;150(7):1377-8. No abstract available. PMID 2369237
- [Background] Eysenbach G. The law of attrition. J Med Internet Res. 2005 Mar 31;7(1):e11. doi: 10.2196/jmir.7.1.e11. PMID 15829473

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Internet Reminder Survey: Treatment phase is 12 months. During the intervention, each subject will receive fluocinonide 0.05% ointment, a standard treatment for psoriasis. If their psoriasis could be suitably treated with fluocinonide, then they will be asked to participate in the study. At the initial study visit, fluocinonide will be dispensed in a small jar with a MEMS® electronic monitoring cap attached. Subjects will be asked to apply the medication twice daily. They will be asked to the entire affected area, excluding face and genitals. Subjects will be instructed to apply the smallest amount of study medication sufficient to cover the affected areas. At the end of the treatment phase, subjects will have a feedback session with specific results of adherence behavior revealed. They will receive weekly surveys via internet to complete.
  Internet Survey
  fluocinonide 0.05% ointment
- Standard of Care, no Internet Survey: Standard treatment for psoriasis. If it is felt that their psoriasis could be suitably treated with fluocinonide, then they will be asked to participate in the study. At the initial study visit, fluocinonide will be dispensed to the subjects in a small jar with a MEMS® electronic monitoring cap attached. Subjects will be asked to apply the medication twice daily. All subjects will be assigned to treatment with topical fluocinonide to the entire affected area, excluding face and genitals. Subjects will be instructed to apply the smallest amount of study medication sufficient to cover the affected areas. At the end of the treatment phase, subjects will have a feedback session with specific results of adherence behavior revealed.
  fluocinonide 0.05% ointment
Period: Overall Study
Arm/Group | Intervention - Internet Reminder Survey | Standard of Care, no Internet Survey
Started | 20 | 20
Completed | 11 | 9
Not Completed | 9 | 11
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Other | 1 | 3
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Population: Description of participants that completed study
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Internet Reminder Survey | Standard of Care, no Internet Survey | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Full Range); unit: years] | 64.81 [50 to 77] | 58.67 [31 to 83] | 62.05 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Measured MEMS Adherence- Number of Days With a Correct Number of Doses Taken
Description: Number of days patients adhered to the treatment is reported. All subjects receive the MEMs caps on their medication and it is reported by the "number" of days that the "dosage" was taken correctly, either with or without internet reminder survey intervention.
  number of days with a correct number of doses taken
Time Frame: up to 12 months
Measure: Mean (Full Range); unit: Days
Arm/Group | Intervention - Internet Reminder Survey | Standard of Care, no Internet Survey
Number analyzed (Participants) | 11 | 9
Days | 15.14 [0.27 to 33.42] | 20.22 [3.125 to 53.3]

2. Secondary Outcome: Mean of Days Per Week Medication Was Taken - Internet Survey
Description: The average number of days per week that participants reported taking the medication in the internet survey
Time Frame: up to 12 months
Population: Includes all participants randomized to this arm. Because the other arm has no internet reminder, there will only be one arm reported for this measure.
Measure: Mean (Full Range); unit: days per week
Arm/Group | Intervention - Internet Reminder Survey
Number analyzed (Participants) | 20
days per week | 5.38 [0 to 6.98]

3. Secondary Outcome: Disease Severity With PASI
Description: Psoriasis Area and Severity Index (PASI): The Psoriasis Area and Severity Index is commonly used in clinical trials as a granular measure of disease severity. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). It is weighted for area in each of the four body regions and scores erythema, induration and desquamation on an overall scale from 0-72. Treatment success is defined as a 75% reduction in PASI score from baseline value.
Time Frame: baseline and 12 months
Population: Data not collected on all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Internet Reminder Survey | Standard of Care, no Internet Survey
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 6.0 (4.64) | 4.31 (2.96)
  month 12: number analyzed (Participants) | 11 | 17
  month 12 | 3.41 (2.16) | 2.94 (2.91)

4. Secondary Outcome: Disease Severity With IGA Assessment
Description: Investigator's Global Assessment (IGA): Similar to assessment performed in clinical practice, based on a 6-point scale from 0 (completely clear) to 5 (very severe). Treatment success is defined as score of 0 or 1 (clear or almost clear).
Time Frame: baseline and 12 months
Population: data not collected in all participants at month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Internet Reminder Survey | Standard of Care, no Internet Survey
Number analyzed (Participants) | 20 | 20
score on a scale
  baseline | 2.6 (.6) | 2.5 (.61)
  month 12: number analyzed (Participants) | 11 | 9
  month 12 | 2.5 (.52) | 2.3 (.5)

ADVERSE EVENTS:
Time Frame: up to 12 months
Arm/Group | Intervention - Internet Reminder Survey | Standard of Care, no Internet Survey
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention - Internet Reminder Survey (N=20) | Standard of Care, no Internet Survey (N=20)
Fungal Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Fungal infection
Burning Sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Burning sensation where drug is applied

LIMITATIONS AND CAVEATS:
A limitation is we did not have continuous measure of disease severity and could not fully assess how much any changes in disease severity affected subjects' use of medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No